CLINICAL TRIAL: NCT07004348
Title: Animation-based Storytelling Education in Relation to Moral Development in 8-12 Year Olds With Dementia-affected Caregivers
Acronym: dementia care
Status: Completed | Type: Observational
Sponsor: Northumbria University (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Frank Lai, Assistant Professor, Northumbria University
Other Study IDs: Northumbria
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Dementia
Keywords: young people; caregivers
MeSH Terms: conditions — Dementia | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Animation group and wait-list group: Animation group will receive 4 sessions of animation as education media as intervention. Wait list group will receive the conventional session of education
  Interventions: Other: Animation group will receive 4 sessions of animation as education media as intervention.

INTERVENTIONS:
Other: Animation group will receive 4 sessions of animation as education media as intervention. — Wait list group will receive the conventional session of education

SUMMARY:
This retrospective, single-blind, parallel group study investigates the impact of animation-based storytelling influence moral development in 8-12 year olds with dementia-affected caregivers.

DETAILED DESCRIPTION:
With the measure of moral reasoning and empathy-related traits to investigate the impact of animation-based storytelling influence moral development in 8-12 year olds with dementia-affected caregivers.

ELIGIBILITY:
Inclusion Criteria:

* full time students in public education. Live with family members who have dementia. Can keep attention for a 15-min animation

Exclusion Criteria:

* any major neurological illness

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: young people in the community
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
The Chinese Prosocial Reasoning Objective Measure (PROM) was used to assess children's moral reasoning. The PROM presents five stories and asks participants to rate the importance of various reasons for helping or not helping in these ethical dilemmas sc | baseline and 1 week after intervention
  The Chinese Prosocial Reasoning Objective Measure (PROM) was used to assess children's moral reasoning. The PROM presents five stories and asks participants to rate the importance of various reasons for helping or not helping in these ethical dilemmas scenarios.

SECONDARY OUTCOMES:
The Chinese interpersonal reactivity index(C-IRI) | baseline and 2 weeks after the intervention
  The Chinese interpersonal reactivity index(C-IRI) is a 21-item self- reported questionnaire measuring empathy-related responses and it has three subscales of personal distress, empathy, and fantasy scale

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lai, Phd, Principal Investigator — The Northumbria University
Locations (1):
- Northumbria University, Newcastle, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Statistical Analysis Plan: PROM link — https://livenorthumbriaac-my.sharepoint.com/:w:/g/personal/frank_lai_northumbria_ac_uk/EbKJJ3cbnk5Ikr-NpppTxHoBmGuJLYpePT6qQ1ZnXA4P-w?e=ZZuX7U